CLINICAL TRIAL: NCT02538887
Title: Use of a Supplemental Radiofrequency Detection System Subsequent to Manual Counting of Vaginal Textiles Following Vaginal Birth: A Prospective Effectiveness and Efficiency Study For Sponge Tracking
Brief Title: Use of a Supplemental Radiofrequency Detection System Subsequent to Manual Counting of Vaginal Textiles Following Vaginal Birth
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor dissolved before study started
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: HSC-MS-15-0535
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Gossyphiboma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Radio Frequency Surgical Detection
  Interventions: Device: Radio Frequency Surgical Detection

INTERVENTIONS:
Device: Radio Frequency Surgical Detection

SUMMARY:
The purpose of this study is to evaluate the FDA-approved Radio Frequency Surgical Detection System (RFDS) as a non-radiological means to ease the process of detecting retained sponges and reconciling sponge counts in the labor and delivery room (following vaginal birth).

DETAILED DESCRIPTION:
This study proposes to evaluate the FDA-approved Radio Frequency Surgical Detection System (RFDS) as a non-radiological means to ease the process of detecting retained sponges and reconciling sponge counts in the labor and delivery room (following vaginal birth). It would not replace any of the current standard-of-care safety mechanisms already in place at the study site to prevent retained sponges. All safeguards remain enforced: counting, visual inspection, and x-rays if indicated by standard protocol. The system being studied involves the surgeon scanning the subject's vaginal area using a spherical device placed 1cm above the symphysis pubis. This static scan will serve to detect any retained cotton textiles within the vaginal cavity after birth. This Verisphere, a reusable device, is encased in a sterile sheath during use. It does not come into direct contact with the subject's vagina, but hovers above the pelvic/vaginal region. If any radio-frequency tagged sponges remain inside the subject, a signal alerts the surgical team to remove them. The visible console displays a confirmation code once the scan is complete. This confirmation code is kept as part of the medical record once absence of retained textiles is confirmed. Once the provider is assured there is no retained item, the same device may be used to scan trash receptacles to locate a missing textile if the pre- and post-delivery sponge/gauze count remains incongruent. This alleviates the need for the assistant personnel to manually "dig" through soiled materials for sponge localization.

ELIGIBILITY:
Inclusion Criteria:

* Adults only, 18 years or older
* Admitted as inpatients to labor and delivery; patients must be in anticipation of vaginal delivery

Exclusion Criteria:

* Urgent or emergent admissions under the influence of preoperative medication, drugs or alcohol.
* Age less than 18 years,
* The patient does not understand English well enough to adequately understand the study.
* Hesitancy of the patient to participate or family reluctance based on the study doctor's opinion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be inpatients at UTHealth/Memorial Hermann Hospital (and affiliates) who are awaiting vaginal birth. Subjects will be identified upon admittance to Labor and Delivery triage.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Estimated); Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients for whom surgical sponge counts can't be reconciled | at the time of radio frequency surgical detection
Number of patients for whom an X-ray was required | at the time of radio frequency surgical detection

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Byrd, MD, Principal Investigator — The University of Texas Health Science Center, Houston